CLINICAL TRIAL: NCT00502580
Title: Evaluation of a Multispectral Vision Enhancement System for Assessment of Oral Mucosal Lesions
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0684
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Oral Cancer
Keywords: Oral Cancer; Multispectral Digital Microscope; Multispectral Digital Imaging; Interview; MDM
MeSH Terms: conditions — Mouth Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pictures of suspicious and normal oral cavity lesions along with small sample of oral lesion (2-4 mm each, the size of a small eraser) will be removed or biopsied from the areas imaged.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with lesions of the oral cavity mucosa.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview taking about 10 minutes to complete.

SUMMARY:
To obtain data to evaluate whether multispectral digital imaging can assist clinicians to screen for premalignant lesions in the oral cavity. Our system will illuminate tissue with monochromatic light to excite fluorescence, and polarized white light to generate reflectance, exposing abnormalities for real time, clinical diagnosis.

Primary Objectives:

1. To compare fluorescence images of oral mucosa lesions, obtained at 350 nm, 380 nm, 400 nm, and 450 nm excitation, to standard white light images and pathologic analysis of biopsied tissue.
2. To compare reflectance images of oral mucosa lesion, obtained using broadband polarized light, to standard white light images and pathologic analysis of biopsied tissue.
3. To develop algorithms to discriminate between normal and abnormal tissue
4. To analyze images to determine which type of optical information (or combination thereof) yields the most diagnostically useful data

DETAILED DESCRIPTION:
All tissue and cells are made of tiny particles that give off small amounts of light. This light is called fluorescence. Scientists have learned that cancerous cells and normal cells give off different amounts and different types of fluorescence. Scientists need to better understand whether fluorescence from the oral cavity (mouth) can be used to tell which cells are abnormal. This information can help doctors detect pre-cancers.

In order to better understand fluorescence, researchers at the Optical Spectroscopy and Imaging Lab, Department of Bioengineering, Rice University have developed an instrument that can collect and analyze fluorescence without surgically removing any tissue or touching the tissue. This instrument takes pictures of oral cavity fluorescence through a microscope. The instrument also takes regular live pictures. Scientists hope to study the pictures to better understand the differences in fluorescence from normal and abnormal cells. The instrument is a standard medical microscope similar to ones used by doctors in their offices to examine people's ears. Researchers have attached a special light source to the microscope that provides different colors of light. In addition, the microscope has a digital camera attached to it so that the researchers can record what they see with the different light colors.

In this study, a clinician will use the instrument to take pictures of suspicious and normal oral cavity lesions. A small sample of the oral lesion (2-4 mm each, the size of a small eraser) will be removed or biopsied from the areas that are imaged. A portion of both the suspicious and normal areas will be taken to pathology for evaluation. The biopsy from the normal appearing area is a biopsy that is additional to those you will receive as part of your standard of care. Each participant will have 2-4 biopsies performed, depending upon how many areas the examiner feels may be suspicious. Most people who take part in this study will be having surgery to remove lesions in the oral cavity anyway, so the biopsies will be performed at the time of surgery. For those participants who are not scheduled to have surgery, the biopsies will be performed under local anesthesia in the clinic.

All data will be numerically coded to ensure your confidentiality.

In addition to the pictures taken and the biopsy, a brief interview will be performed by the clinical research staff to discuss possible past local therapies and your personal history of tobacco and alcohol use. The interview should take about 10 minutes to complete.

You will not be told of any of the experimental findings. Information confirming the diagnosis will be made available to your treating physician. After this visit and tissue collection, your participation in this study will be complete.

This is an investigational study. A total of 45 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with lesions of the oral cavity mucosa or suspicious for malignancy or premalignancy.
2. Subjects with the ability and willingness to sign an informed consent and authorization.
3. Subjects who develop new lesions or alterations in long-standing lesions are eligible, but not required, for re-examination with informed consent.

Exclusion Criteria:

1. Persons who are medically unfit to undergo superficial punch biopsies of oral mucosa.
2. Persons under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lesions of the oral cavity mucosa.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2005-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Evaluate new imaging technology, MDM (Multispectral Digital Microscope), as a tool for early diagnosis of oral neoplasia | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Gillenwater, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org